CLINICAL TRIAL: NCT06851572
Title: Prevalence of Late Xerostomia and Hyposalivation with Associated Risk Factors in Survivors of Head and Neck Cancer After Radiotherapy: a Multi-centric Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Other Study IDs: HAM00221
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Radiotherapy Side Effect; Xerostomia Due to Radiotherapy; Xerostomia Due to Radiotherapy (Disorder)
Keywords: dry mouth, xerostomia, hyposalivation, head and neck, cancer, radiotherapy.
MeSH Terms: conditions — Radiation Injuries; Xerostomia; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study titled "Prevalence of Late Xerostomia and Hyposalivation with Associated Risk Factors in Survivors of Head and Neck Cancer After Radiotherapy" is a multi-centric cross-sectional study conducted in Egypt. It aims to assess the prevalence of late-onset xerostomia (dry mouth) and hyposalivation in survivors of head and neck cancer (HNC) who have undergone radiotherapy. Given the widespread use of radiotherapy as a treatment for HNC, its long-term side effects-especially on salivary gland function-are a major concern for patient quality of life.

The study includes 260 participants who have completed curative radiotherapy at least one year prior, with or without chemotherapy. Patients were selected from multiple centers, and eligibility criteria required them to be at least 18 years old. Those with recurrent or secondary malignancies were excluded. The researchers hypothesized that high doses of radiation administered to the salivary glands would lead to a high prevalence of xerostomia, and that concomitant chemotherapy might further exacerbate this condition.

To evaluate xerostomia, both subjective and objective assessments were conducted. The Summated Xerostomia Inventory (SXI), a five-item questionnaire, was used to measure self-reported symptoms of dry mouth. Objective assessments included salivary flow rate measurement, oral dryness indicators, and glandular response to stimulation. Additionally, the MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) was used to assess the impact of xerostomia on daily functioning and quality of life.

The study also examined various risk factors associated with xerostomia, including tumor site, treatment type (radiotherapy alone or with chemotherapy), demographic factors (age, gender, education level), and lifestyle habits (such as smoking status). Smoking history was classified into never smokers, former smokers (quit >6 months before diagnosis), and current smokers (either quit post-diagnosis or continued smoking).

This research is significant as it is one of the first large-scale studies in Egypt to evaluate long-term salivary dysfunction in head and neck cancer survivors. By identifying prevalence rates and contributing factors, the study provides valuable insights for improving patient care and developing better management strategies for individuals suffering from post-radiotherapy xerostomia.

DETAILED DESCRIPTION:
Cancer of the oral cavity, pharynx, and larynx corresponds to approximately 4.6% of all cases of cancer worldwide.[1] In 2018, 834,860 new cases of cancer in these anatomic sites were diagnosed.[1] When anatomic sub-sites are analyzed, the incidence of cancer of the mouth and oropharynx is higher, followed by cancer of the larynx and hypopharynx.[2] Due to demographic changes, the number of cases of lip, mouth, and pharyngeal cancer is expected to increase by 62%, reaching 856,000 cases annually by 2035.[3] Radiotherapy (RT) is widely employed in the treatment of head and neck cancer used as primary therapy, adjunct therapy to surgery, with concomitant chemotherapy (CT) or as palliative treatment. High doses of RT can negatively affect the soft and hard tissues of the oral cavity.[4] Patients with head and neck cancer are generally irradiated with high doses (50 to 70 Gy),[5] which side-effects include xerostomia, trismus, and dysphagia; in hard tissues, the effects may be osteoradionecrosis and radiation caries all of which have a late-onset.[4] One of the main problems resulting from radiotherapy in the head and neck region is the damage to glandular tissues, reducing the salivary flow.[6] Xerostomia occurs due to cell death and fibrosis of the glandular tissue caused by radiotherapy, leading to a sensation of dry mouth (xerostomia).[7] Some studies suggest a significant increase in late onset xerostomia in patients treated with concomitant chemotherapy and radiotherapy,[8] whereas other authors state that there is no strong evidence of the additive effect of chemotherapy concomitant to radiotherapy on hypofunction of the salivary glands.[9] In a systematic review, Jensen, et al.[9] (2010) found divergences in the literature regarding hyposalivation and xerostomia. According to some authors, the term xerostomia is often used as a synonym of hyposalivation, when it should only be used to indicate the perception of dry mouth reported by the patient.[3] Due to this common late effect in patients irradiated in head and neck and the influence on their quality of life, studies bringing new information to the field are necessary. Therefore, this study evaluates the prevalence and factors associated with late xerostomia based on the stimulated salivary flow rate in patients treated with Intensity-modulated radiation therapy (IMRT) with or without concomitant chemotherapy for the treatment of cancer of the oral cavity, oropharynx, hypopharynx, or larynx. We hypothesize that a high prevalence would be found caused by high doses of radiation in the salivary glands and also influenced by the type of therapy used in this region in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck Cancer (HNC) Survivors

Must have completed curative radiotherapy for HNC at least 1 year prior (with or without chemotherapy).

Aged 18 years or older. Willing to provide informed consent and undergo dry mouth assessment.

Exclusion Criteria:

* Recurrent or Secondary Malignancies

Patients with recurrent HNC or a new secondary primary cancer before survey administration.

❌ Severe Comorbid Conditions

Any systemic disease or medical condition that significantly impacts salivary function (e.g., Sjögren's syndrome, uncontrolled diabetes, autoimmune diseases).

❌ Recent Radiotherapy or Ongoing Cancer Treatment

Patients who underwent radiation within the past year. Those receiving active cancer treatment during the study period.

❌ Non-Consent or Cognitive Impairment

Patients who are unwilling to participate or unable to complete questionnaires due to cognitive dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on long-term survivors of head and neck cancer (HNC) who have undergone curative radiotherapy with or without chemotherapy. The population includes both male and female patients who have completed their treatment at least one year prior to participation.
  Patients will be recruited from multiple medical centers, ensuring a diverse and representative sample of HNC survivors. The study aims to assess the prevalence of late-onset xerostomia and hyposalivation, along with associated risk factors such as treatment type, tumor characteristics, smoking status, and sociodemographic variables.
  The study specifically targets individuals aged 18 years or older, with no recurrent or secondary primary malignancies, and who are willing to participate in subjective and objective assessments of salivary gland dysfunction.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Summated Xerostomia Inventory (SXI) | single point "Baseline"
  the Summated Xerostomia Inventory (SXI), which consists of five subjective statements related to dry mouth symptoms. Each statement is scored from 1 (never) to 3 (often), with a maximum score of 15, indicating severe xerostomia.

SECONDARY OUTCOMES:
unstimulated salivary flow rate | single point "Baseline"
  Measured using unstimulated salivary flow rate collected over 5 minutes and expressed in mL/min. Patients will be classified as having normal, reduced, or absent salivary flow.
Quality of Life (QoL) | single point "Baseline"
  Assessed using the MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN), a 28-item questionnaire measuring symptom severity and daily life interference on a 0-10 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided